CLINICAL TRIAL: NCT03839407
Title: The Impact of the MUSE Meditation Device on Perceived Stress, Anxiety, Affect, and Burnout Among Student Registered Nurse Anesthetists
Brief Title: The Impact of the MUSE Meditation Device on Student Registered Nurse Anesthetists
Acronym: MUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diana J. Kelm (Other)
Responsible Party: Sponsor-Investigator, Diana J. Kelm, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-011173
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Stress; Anxiety; Affect; Burnout, Professional
MeSH Terms: conditions — Anxiety Disorders; Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MUSE device Class 21 (Experimental): Participants will utilize the MUSE device for 12 weeks during the intervention period.
  Interventions: Device: MUSE Meditation Device
- No MUSE device Class 21 (No Intervention): Participants will not utilize the MUSE device for 12 weeks during the non-intervention period.
- MUSE device Class 22 (Experimental): Participants will utilize the MUSE device for 12 weeks during the intervention period.
  Interventions: Device: MUSE Meditation Device
- No MUSE device Class 22 (No Intervention): Participants will not utilize the MUSE device for 12 weeks during the non-intervention period.

INTERVENTIONS:
Device: MUSE Meditation Device — The MUSE Meditation Device guides users in mindful meditation using real-time feedback on brain wave activity.
  Arms: MUSE device Class 21; MUSE device Class 22

SUMMARY:
The question this study is designed to answer is whether or not the use of a MUSE Meditation Device lowers student registered nurse anesthetist's perception of stress, anxiety, and burnout within the Mayo Clinic Doctorate of Nurse Anesthesia Practice Program.

ELIGIBILITY:
Inclusion Criteria:

* Student Registered Nurse Anesthetists at Mayo Clinic in the class of 2021 and 2022.

Exclusion Criteria:

* Student Registered Nurse Anesthetists at Mayo Clinic who are not in the class of 2021 and 2022.

Ages: 24 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Change in Stress, as measured by the Perceived Stress Scale-10 | baseline and 3, 6, and 12 months
  Scores range from 0 to 40 with 0 indicating no stress and a higher score indicating greater stress.

SECONDARY OUTCOMES:
Change in Anxiety, as measured by the Generalized Anxiety Disorder Scale-7 | baseline and 3, 6, and 12 months
  Scores range from 0 to 21 with 0 indicating no anxiety and a higher score indicating greater anxiety.
Change in Affect, as measured by the Positive and Negative Affect Scale | baseline and 3, 6, and 12 months
  Scores range from 10-50 within positive and negative scales. The higher the score, the higher the positive or negative affect.
Change in Burnout, as measured by the Maslach Burnout Inventory-2 | baseline and 3, 6, and 12 months
  A two question survey asking the participant burnout questions within the workplace.
Change in Self-Perceived Medical Error, as measured by a single question. | 3 & 6 months
  A single yes or no question asking if participant felt they made any medical errors

CONTACTS AND LOCATIONS:
Overall Officials: Diana Kelm, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials